CLINICAL TRIAL: NCT01707147
Title: A Regulatory Requirement Non Interventional Study to Monitor the Safety and Effectiveness of Trajenta (Linagliptin, 5 mg, q.d) in Korean Patients With Type 2 Diabetes Mellitus(SELINA Study)
Brief Title: A Non Interventional Study to Monitor the Safety and Effectiveness of Trajenta (Linagliptin, 5 mg, q.d) in Korean Patients With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1218.104
Record Dates: First submitted 2012-10-01; First posted 2012-10-16 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with Type 2 Diabetes Mellitus
  Interventions: Drug: Trajenta tablet

INTERVENTIONS:
Drug: Trajenta tablet — Linagliptin

SUMMARY:
The aim of this study is to monitor safety and efficacy of treatment with linagliptin in Korean patients with type 2 diabetes mellitus in routine clinical settings.

DETAILED DESCRIPTION:
Study Design:

Post Marketing study- Observational study

ELIGIBILITY:
Inclusion criteria:

Patients who have been started on Trajenta in accordance with the approved label in Korea Patients who have signed on the data release consent form

Exclusion criteria:

Patients with previous exposure to Trajenta and current participation in clinical trials

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients with T2DM
Sampling Method: Probability Sample
Enrollment: 3219 (Actual)
Dates: Start 2012-11-16 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Multiple Locations, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A regulatory requirement prospective, non-interventional, open-label, multi-centre national study to monitor the safety and effectiveness of Trajenta (Linagliptin, 5 milligram (mg), once daily) in Korean patients with type 2 diabetes mellitus
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended a specialist sites which ensured that they met all strictly implemented inclusion/exclusion criteria. Patients were not to be entered to trial if any one of the specific entry criteria was violated.
Groups:
- Trajenta (Linagliptin) 5 mg: Patients with type 2 diabetes mellitus were administered with Trajenta (Linagliptin) 5 mg once daily orally.
Period: Overall Study
Arm/Group | Trajenta (Linagliptin) 5 mg
Started (Number of patients in case report form (CRF) collection) | 3219
Completed (Number of patients in safety analysis set) | 3119
Not Completed | 100
Not completed — Administered Trajenta prior to contract | 5
Not completed — Patients who have not taken Trajenta | 1
Not completed — Follow-up failure | 17
Not completed — Violated inclusion/exclusion criteria | 77

BASELINE CHARACTERISTICS:
Population: Safety analysis set: This analysis set included all patients who were administrated Trajenta at least once, except patients violating inclusion/exclusion criteria, dosage administration or lost to follow up.
Arm/Group | Trajenta (Linagliptin) 5 mg
Number analyzed (Participants) | 3119
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Number of patients in safety analysis set
  Years | 61.24 (11.95)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number of patients in safety analysis set
  Participants
    Female | 1450
    Male | 1669
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — All patients in the safety set were Korean because this was an inclusion criteria Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Incidence of Adverse Events Who Had Taken at Least One Dose of Trajenta
Description: Percentage of patients with incidence of any adverse events who had taken at least one dose of Trajenta.
Time Frame: Up to 26 weeks (long-term surveillance)
Population: as for baseline characteristics
Measure: Number; unit: Percentage of patients
Arm/Group | Trajenta (Linagliptin) 5 mg
Number analyzed (Participants) | 3119
Percentage of patients | 7.69

2. Secondary Outcome: Change From Baseline After 24 Weeks in Glycosylated Hemoglobin (HbA1c)
Description: Change from baseline after 24 weeks in Glycosylated Hemoglobin (HbA1c).
Time Frame: Baseline and Week 24
Population: Effectiveness analysis set: This set includes all patients of the safety analysis set for whom HbA1c values were measured at both baseline and after drug administration.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Trajenta (Linagliptin) 5 mg
Number analyzed (Participants) | 2171
Percentage of HbA1c
  Before drug administration | 7.98 (1.51)
  After drug administration | 7.21 (1.22)
Statistical Analysis 1: Comparison: Trajenta (Linagliptin) 5 mg; Test type: Other; p < 0.0001, Paired t-test; Mean Difference (Final Values) = -0.77, 95% CI 2-sided [-0.83 to -0.71], Standard Deviation 1.50 — p-value of paired t-test for change from baseline is presented. 95% confidence interval for the mean was calculated using t-distribution

3. Secondary Outcome: Percentage of Patients With Occurrence of Treat to Target Effectiveness Response, That is HbA1c Under Treatment of < 6.5% After 24 Weeks of Treatment
Description: Percentage of patients with occurrence of treat to target effectiveness response, that is HbA1c under treatment of < 6.5% after 24 weeks of treatment.
Time Frame: 24 Weeks
Population: Effectiveness analysis set
Measure: Number; unit: Percentage of patients
Arm/Group | Trajenta (Linagliptin) 5 mg
Number analyzed (Participants) | 2171
Percentage of patients | 26.02

4. Secondary Outcome: Percentage of Patients With Occurrence of Relative Effectiveness Response (HbA1c Lowering by at Least 0.5% After 24 Weeks of Treatment)
Description: Percentage of patients with occurrence of relative effectiveness response (HbA1c lowering by at least 0.5% after 24 weeks of treatment).
Time Frame: 24 Weeks
Population: Effectiveness analysis set
Measure: Number; unit: Percentage of patients
Arm/Group | Trajenta (Linagliptin) 5 mg
Number analyzed (Participants) | 2171
Percentage of patients | 57.30

5. Secondary Outcome: Change From Baseline After 24 Weeks in Fasting Plasma Glucose (FPG)
Description: Change from baseline after 24 weeks in fasting plasma glucose (FPG).
Time Frame: Baseline and Week 24
Population: Effectiveness analysis set: the patients with the data available for FPG
Measure: Mean (Standard Deviation); unit: Milligrams per Deciliter
Arm/Group | Trajenta (Linagliptin) 5 mg
Number analyzed (Participants) | 2171
Milligrams per Deciliter
  Before drug administration: number analyzed (Participants) | 1863
  Before drug administration | 161.19 (55.38)
  After drug administration: number analyzed (Participants) | 1820
  After drug administration | 143.51 (46.76)
Statistical Analysis 1: Comparison: Trajenta (Linagliptin) 5 mg; Test type: Other; p < 0.0001, Paired t-test; Mean Difference (Final Values) = -18.05, 95% CI 2-sided [-20.98 to -15.12], Standard Deviation 61.84 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: From the entire surveillance period until re-examination period, up to 6 years.
Arm/Group | Trajenta (Linagliptin) 5 mg
All-Cause Mortality (participants affected / at risk) | 2/3119
Serious Adverse Events (participants affected / at risk) | 49/3119
Other Adverse Events (participants affected / at risk) | 0/3119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trajenta (Linagliptin) 5 mg (N=3119)
Constipation (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Herpes zoster (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Vestibular neuronitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cerebral infarction (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Dementia Alzheimer's type (Nervous system disorders) | 1
Chest pain (General disorders) | 1
Pyrexia (General disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 1
Death (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1
Pneumoconiosis (Injury, poisoning and procedural complications) | 1
Cardiac failure congestive (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Diabetic retinopathy (Eye disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
End stage renal disease (Renal and urinary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholangitis (Hepatobiliary disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Renal transplant failure (Immune system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT01707147/SAP_000.pdf
  • Study Protocol (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/47/NCT01707147/Prot_001.pdf